CLINICAL TRIAL: NCT02728089
Title: A Multicenter, Open-label, Noncomparative, Japanese Phase III Study to Assess the Efficacy and Safety of Ceftolozane/Tazobactam (MK-7625A) in Japanese Patients With Uncomplicated Pyelonephritis and Complicated Urinary Tract Infection
Brief Title: Study of Ceftolozane/Tazobactam (MK-7625A) in Japanese Participants With Uncomplicated Pyelonephritis and Complicated Urinary Tract Infection (MK-7625A-014)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-014; MK-7625A-014 (Other: Merck Registration Number); 163276 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Urinary Tract Infection (UTI); Complicated Urinary Tract Infection; Pyelonephritis; Uncomplicated Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — ceftolozane; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-7625A (Experimental): MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) administered as an intravenous (IV) infusion every 8 hours for 7 days. The dose may be reduced to 750 mg (ceftolozane 500 mg/tazobactam 250 mg) for participants with a creatinine clearance (CrCl) of 30-50 mL/min.
  Interventions: Drug: MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g)

INTERVENTIONS:
Drug: MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) — MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) administered as an intravenous (IV) infusion

SUMMARY:
This is a Phase 3, multi-site, non-randomized, open-label study evaluating the safety and efficacy of MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) for the treatment of complicated urinary tract infection (cUTI) including pyelonephritis (uncomplicated or complicated pyelonephritis and complicated lower urinary tract infection) in Japanese participants. Efficacy will be primarily assessed by microbiological response defined as eradication of the baseline pathogen or pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males or females who need hospitalization
* Clinical signs and/or symptoms of urinary tract infection (UTI) at screening visit, either one of the following:

  * Pyelonephritis (uncomplicated or complicated)
  * Complicated lower UTI (cUTI)
* Has a pretreatment baseline urine culture specimen obtained within 24 hours of start of study drug
* Requires IV antibacterial therapy for the treatment of the presumed UTI
* Female participants of child bearing potential must not be pregnant (negative human chorionic gonadotropin test) or breastfeeding and must agree to use adequate contraception for the duration of the study and up to 35 days after the last dose of study drug
* Male participants must agree to use adequate contraception for the duration of the study and up to 75 days after the last dose of study drug

Exclusion Criteria:

* Has a history of recent or recurrent Gram-positive organism UTI suggesting colonization, or participant with UTI that shows or suspects the presence of a Gram-positive organism only
* Has a history of any moderate or severe hypersensitivity or allergic reaction to any Beta-lactam antibacterial including cephalosporins, carbapenems and penicillins, or tazobactam
* Has a concomitant infection at the time of randomization, which requires non-study systemic antibacterial therapy in addition to study drug with the exception of an antibacterial with Gram-positive activity only (vancomycin, linezolid, daptomycin and teicoplanin)
* Is receiving probenecid
* Is currently receiving bladder infusions with topical urinary antiseptics or antibacterial agents
* Has received any amount of potentially therapeutic antibacterial therapy after collection of the pretreatment baseline urine culture and before administration of the first dose of study drug.
* Has received any dose of a potentially therapeutic antibacterial agent for the treatment of the current UTI within 48 hours before the pretreatment baseline urine is obtained
* Intractable urinary infection at baseline that would require more than 7 days of study drug
* Has complete, permanent obstruction of the urinary tract.
* Has confirmed fungal urinary tract infection at time of randomization (with ≥ 10^3 fungal colony forming units /mL)
* Has permanent indwelling bladder catheter or urinary stent including nephrostomy
* Has suspected or confirmed perinephric or intrarenal abscess
* Has suspected or confirmed prostatitis, urethritis, or epididymitis
* Has ileal loop or known vesico-ureteral reflux
* Severe impairment of renal function including an estimated CrCl < 30 mL/min, requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (< 20 mL/hr urine output over 24 hours)
* Has urinary catheter that is not scheduled to be removed before the end of therapy
* Has any rapidly progressing disease or immediately life-threatening illness including acute hepatic failure, respiratory failure, and septic shock
* Has an immunocompromising condition (i.e., AIDS, hematological malignancy, or bone marrow transplantation, or immunosuppressive therapy) or is receiving ≥ 40 mg of prednisone per day administered continuously for > 14 days prior to study start
* Has participated in any clinical study of an investigational product within 30 days prior to the first dose of study drug
* Has previously participated in any study of ceftolozane or MK-7625A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Arakawa S, Kawahara K, Kawahara M, Yasuda M, Fujimoto G, Sato A, Yokokawa R, Yoshinari T, Rhee EG, Aoyama N. The efficacy and safety of tazobactam/ceftolozane in Japanese patients with uncomplicated pyelonephritis and complicated urinary tract infection. J Infect Chemother. 2019 Feb;25(2):104-110. doi: 10.1016/j.jiac.2018.10.009. Epub 2018 Nov 9. PMID 30420153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-7625A
Started | 115
Treated | 114
Completed | 112
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MK-7625A
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 115
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Microbiological Response of Eradication at Test of Cure (TOC)
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline at TOC (14 days post first dose). Microbiological outcome was classified as "eradication", "persistence" or "indeterminate." A successful microbiological response was "eradication" which was defined as urine culture showed all uropathogens found at baseline at ≥10^5 colony-forming unit (CFU)/mL were reduced to <10^4 CFU/mL. If the outcome for any uropathogen was" persistence" (CFU/mL not reduced the result was classified as unsuccessful. Participants with responses reported as "indeterminate" were excluded.
Time Frame: Day 14 (14 days post first dose of study drug)
Population: All participants who received at least 1 dose of study drug, had at least 1 acceptable causative uropathogen at baseline, adhered to study procedures, had a clinical response at the visit of interest within specified visit window, had an appropriately collected urine culture specimen and interpretable urine culture result at the visit of interest.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 88
Percentage of participants | 80.7 [70.9 to 88.3]

2. Primary Outcome: Percentage of Participants Who Report 1 or More Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized.
Time Frame: Up to 42 days post first dose of study drug
Population: All participants who received at least 1 dose of study treatment and had follow-up data for endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 114
Percentage of participants | 58.8 [49.2 to 67.9]

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not considered related to the medicinal product. The percentage of participants that had study drug discontinued during the study due to an AE was summarized.
Time Frame: Up to 7 days after the first dose of study drug
Population: All participants who received at least 1 dose of study treatment and had follow-up data for endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 114
Percentage of participants | 1.8 [0.2 to 6.2]

4. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication at End Of Therapy (EOT)
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline at EOT (7 days post first dose of study drug). Microbiological outcome was classified as "eradication", "persistence" or "indeterminate." A successful microbiological response was "eradication" which was defined as urine culture showed all uropathogens found at baseline at ≥10^5 colony-forming unit (CFU)/mL were reduced to <10^4 CFU/mL. If the outcome for any uropathogen was" persistence" (CFU/mL not reduced the result was classified as unsuccessful. Participants with responses reported as "indeterminate" were excluded.
Time Frame: Day 7 (7 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 87
Percentage of participants | 100.0 [95.8 to 100.0]

5. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication at Late Follow-up (LFU)
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline at LFU (42 days post first dose of study drug). Microbiological outcome was classified as "eradication", "persistence" or "indeterminate." A successful microbiological response was "eradication" which was defined as urine culture showed all uropathogens found at baseline at ≥10^5 colony-forming unit (CFU)/mL were reduced to <10^4 CFU/mL. If the outcome for any uropathogen was" persistence" (CFU/mL not reduced the result was classified as unsuccessful. Participants with responses reported as "indeterminate" were excluded.
Time Frame: Day 42 (42 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 82
Percentage of participants | 61.0 [49.6 to 71.6]

6. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at TOC
Description: The Investigator classified clinical outcome as "clinical cure", "clinical failure", or "indeterminate". A favorable clinical response is "clinical cure" defined as complete resolution of, marked improvement in (where clinical improvement was defined as a reduction in severity of all baseline signs and symptoms with worsening of none and with no requirement for additional antibiotic therapy after EOT), or return to pre-infection signs and symptoms and no use of additional or nonstudy antimicrobial therapy for the treatment of the current UTI. Outcomes reported as "indeterminate" were excluded. Percentage of participants with clinical response of clinical cure at TOC was summarized
Time Frame: Day 14 (14 days post first dose of study drug)
Population: All participants who received at least 1 dose of study treatment, had at least 1 acceptable causative uropathogen at baseline, adhered to study procedures and had a clinical response at the visit of interest within the specified visit window. All participants had to have an evaluable clinical outcome; an indeterminate response was excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 89
Percentage of participants | 96.6 [90.5 to 99.3]

7. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at EOT
Description: The Investigator classified clinical outcome as "clinical cure", "clinical failure", or "indeterminate". A favorable clinical response is "clinical cure" defined as complete resolution of, marked improvement in (where clinical improvement was defined as a reduction in severity of all baseline signs and symptoms with worsening of none and with no requirement for additional antibiotic therapy after EOT), or return to pre-infection signs and symptoms and no use of additional or nonstudy antimicrobial therapy for the treatment of the current UTI. Outcomes reported as "indeterminate" were excluded. Percentage of participants with clinical response of clinical cure at EOT was summarized
Time Frame: Day 7 (7 days post first dose of study drug)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 89
Percentage of participants | 97.8 [92.1 to 99.7]

8. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at LFU
Description: The Investigator classified clinical outcome as "clinical cure", "clinical failure", or "indeterminate". A favorable clinical response is "clinical cure" defined as complete resolution of, marked improvement in (where clinical improvement was defined as a reduction in severity of all baseline signs and symptoms with worsening of none and with no requirement for additional antibiotic therapy after EOT), or return to pre-infection signs and symptoms and no use of additional or nonstudy antimicrobial therapy for the treatment of the current UTI. Outcomes reported as "indeterminate" were excluded. Percentage of participants with clinical response of clinical cure at LFU was summarized.
Time Frame: Day 42 (42 days post first dose of study drug)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 87
Percentage of participants | 78.2 [68.0 to 86.3]

9. Secondary Outcome: Percentage of Participants With a Composite Response of Both Eradication and Clinical Cure at TOC
Description: The percentage of participants that met requirements for both eradication and clinical cure at TOC was summarized.
Time Frame: Day 14 (14 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 88
Percentage of participants | 80.7 [70.9 to 88.3]

10. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication, by Pathogen at EOT
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline. Microbiological outcome was classified as "Eradication", "Persistence" or "Indeterminate." A successful microbiological response was "Eradication" which was defined as urine culture showed the specific pathogen found at baseline at ≥10^5 colony-forming unit (CFU)/mL was reduced to <10^4 CFU/mL. If the outcome for any uropathogen was persistence (CFU/mL not reduced the result was classified as a failure. Outcomes reported as "indeterminate" were excluded. The percentage of participants that achieved eradication for each uropathogen at EOT (7 days post first dose of study drug) was summarized.
Time Frame: Day 7 (7 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 87
Percentage of participants
  Enterobacter aerogenes: number analyzed (Participants) | 1
  Enterobacter aerogenes | 100.0 [2.5 to 100.0]
  Escherichia coli: number analyzed (Participants) | 76
  Escherichia coli | 100.0 [95.3 to 100.0]
  Klebsiella pneumoniae: number analyzed (Participants) | 7
  Klebsiella pneumoniae | 100.0 [59.0 to 100.0]
  Proteus mirabilis: number analyzed (Participants) | 2
  Proteus mirabilis | 100.0 [15.8 to 100.0]
  Proteus vulgaris: number analyzed (Participants) | 2
  Proteus vulgaris | 100.0 [15.8 to 100.0]
  Pseudomonas aeruginosa: number analyzed (Participants) | 1
  Pseudomonas aeruginosa | 100.0 [2.5 to 100.0]

11. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication by Pathogen at TOC
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline. Microbiological outcome was classified as "Eradication", "Persistence" or "Indeterminate." A successful microbiological response was "Eradication" which was defined as urine culture showed the specific pathogen found at baseline at ≥10^5 colony-forming unit (CFU)/mL was reduced to <10^4 CFU/mL. If the outcome for any uropathogen was persistence (CFU/mL not reduced), the result was classified as a failure. Outcomes reported as "indeterminate" were excluded. The percentage of participants that achieved eradication for each uropathogen at TOC (14 days post first dose of study drug) was summarized.
Time Frame: Day 14 (14 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 88
Percentage of participants
  Citrobacter koseri: number analyzed (Participants) | 1
  Citrobacter koseri | 100.0 [2.5 to 100.0]
  Enterobacter aerogenes: number analyzed (Participants) | 1
  Enterobacter aerogenes | 100.0 [2.5 to 100.0]
  Escherichia coli: number analyzed (Participants) | 76
  Escherichia coli | 82.9 [72.5 to 90.6]
  Klebsiella pneumoniae: number analyzed (Participants) | 7
  Klebsiella pneumoniae | 42.9 [9.9 to 81.6]
  Proteus mirabilis: number analyzed (Participants) | 3
  Proteus mirabilis | 100.0 [29.2 to 100.0]
  Proteus vulgaris: number analyzed (Participants) | 2
  Proteus vulgaris | 100.0 [15.8 to 100.0]
  Pseudomonas aeruginosa: number analyzed (Participants) | 1
  Pseudomonas aeruginosa | 100.0 [2.5 to 100.0]

12. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication by Pathogen at LFU
Description: The per-pathogen microbiological outcome was determined for each uropathogen isolated at baseline. Microbiological outcome was classified as "Eradication", "Persistence" or "Indeterminate." A successful microbiological response was "Eradication" which was defined as urine culture showed the specific pathogen found at baseline at ≥10^5 colony-forming unit (CFU)/mL was reduced to <10^4 CFU/mL. If the outcome for any uropathogen was persistence (CFU/mL not reduced the result was classified as a failure. Outcomes reported as "indeterminate" were excluded. The percentage of participants that achieved eradication for each uropathogen LFU (42 days post first dose of study drug) was summarized.
  .
Time Frame: Day 42 (42 days post first dose of study drug)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-7625A
Number analyzed (Participants) | 82
Percentage of participants
  Citrobacter koseri: number analyzed (Participants) | 1
  Citrobacter koseri | 100.0 [2.5 to 100.0]
  Enterobacter aerogenes: number analyzed (Participants) | 1
  Enterobacter aerogenes | 100.0 [2.5 to 100.0]
  Escherichia coli: number analyzed (Participants) | 70
  Escherichia coli | 62.9 [50.5 to 74.1]
  Klebsiella pneumoniae: number analyzed (Participants) | 8
  Klebsiella pneumoniae | 37.5 [8.5 to 75.5]
  Proteus mirabilis: number analyzed (Participants) | 3
  Proteus mirabilis | 66.7 [9.4 to 99.2]
  Proteus vulgaris: number analyzed (Participants) | 1
  Proteus vulgaris | 100.0 [2.5 to 100.0]
  Pseudomonas aeruginosa: number analyzed (Participants) | 1
  Pseudomonas aeruginosa | 100.0 [2.5 to 100.0]

ADVERSE EVENTS:
Time Frame: up to 35 post last dose of study drug (up to 42 days total)
Description: All participants that received at least 1 dose of study drug
Arm/Group | MK-7625A
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 13/114
Other Adverse Events (participants affected / at risk) | 26/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7625A (N=114)
Cardiac failure (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 3 (3)
Pyelonephritis chronic (Infections and infestations) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7625A (N=114)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 9 (9)
Alanine aminotransferase increased (Investigations) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02728089/Prot_SAP_000.pdf